CLINICAL TRIAL: NCT01287195
Title: Oral Anti-CD3 for the Treatment of Active Ulcerative Colitis
Brief Title: Oral OKT3 for the Treatment of Active Ulcerative Colitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Scott B. Snapper, M.D., Ph.D., Director, Inflammatory Bowel Disease Research, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009P001448
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-01

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Muromonab-CD3; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral OKT3 (Experimental): Participants with ulcerative colitis will receive Oral OKT3 given with Omeprazole once daily for 30 days.
  Interventions: Drug: Oral OKT3; Drug: Omeprazole

INTERVENTIONS:
Drug: Oral OKT3 — 1 mg or 2 mg Oral OKT3 will be given orally to participants once daily for 30 days
  Other Names: Muromonab CD3; OKT3; anti-CD3
Drug: Omeprazole — 20 mg Omeprazole will be given orally to participants once daily for 30 days
  Other Names: Prilosec

SUMMARY:
This study will assess the safety and efficacy of orally delivered short-term OKT3 in participants with active ulcerative colitis.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic disease of unknown etiology characterized by infiltration of inflammatory cells into the intestinal tract. OKT3 is an approved drug for intravenous use in the treatment of solid-organ transplantation. However, intravenous dosing has been limited by significant toxicities. Data from animal models suggest that antibody recognizing the T3 antigen complex Cluster of Differentiation 3 (anti-CD3) administered via the oral route is effective at treating a variety of autoimmune diseases. No side effects were observed in a recent phase I study of healthy participants receiving oral anti-CD3 monoclonal antibody (mAb).

The objectives of the current study are to assess the safety, immunologic effects and efficacy of short-term oral administration of OKT3 in participants with active ulcerative colitis. OKT3 will be delivered orally as a 1 milligram (mg) or 2 mg dose with Omeprazole 20 mg daily for 30 consecutive days in an open-label pilot trial. Thirty two participants will be screened for a targeted completion of 16 enrolled participants. The participants will be evaluated at baseline, day 1, day 2, week 1, week 3, as well as after completion of therapy at week 5 and 10 after the initiation of treatment. Lab tests will be performed at screening, baseline, day 2, week 1, week 3, week 5 and week 10. Clinical data will be collected at all study visits and via diary entries throughout the study period. A flexible sigmoidoscopy will be done at baseline and at week 5. Stool studies will be performed at screening to rule out infection.

To be eligible for this study, participants must be between the ages of 18 and 65 years and have a history of moderately to severely active UC as defined by a Mayo score of 6 to 12. They may not be taking concurrent biologic or immunomodulator therapy for UC.

ELIGIBILITY:
1.1 Inclusion Criteria

* Ability to provide informed consent
* Age between 18 and 65 years
* Confirmed diagnosis of UC for at least 3 months with the extent defined within the previous year
* Moderate to severe UC as defined by a Mayo score of 6-12
* Concomitant medications: Can be on 5-amino salicylate (5-ASA) medications and stable doses (same dose > 4 weeks) of oral steroids
* Concomitant medications cannot include Infliximab, Adalimumab, Certolizumab or Natalizumab for 4 weeks; rectal steroids, 6-mercaptopurine (6-MP), Azathioprine, Tacrolimus, Methotrexate, Thalidomide, Cellcept for 4 weeks; Theophylline, sulfonylureas, non-steroidal anti-inflammatory drug (NSAIDs) or aspirin for 10 days
* Negative serum pregnancy test within 2 weeks prior to receiving the first dose of study drug in female participants of child-bearing potential
* Female participants of child-bearing potential must be willing to use birth control during the study and for 4 weeks following the last dose of study drug.

1.2 Exclusion Criteria

* Crohn's disease or indeterminate colitis
* Mayo score of <6 (mild UC)
* Hospitalized or exhibiting signs of toxicity (abdominal distension, severe abdominal tenderness, fever, nausea, vomiting, or tachycardia)
* A history of colorectal cancer or colorectal dysplasia
* Pregnant or breastfeeding females or females wishing to become pregnant within the next 6 months or unwilling to use birth control
* Serum creatinine ≥ 2.0 milligrams per deciliter (mg/dL)
* Alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), or direct bilirubin >1.5x normal: elevated indirect bilirubin related to likely Gilbert's disease permissible
* Use of any of the following medications: Azathioprine, 6-MP, Methotrexate, Mycophenolate Mofetil, Tacrolimus, Cyclosporine, Thalidomide, Adalimumab, Infliximab, Certolizumab, Natalizumab, rectal steroids. Theophylline, sulfonylureas, NSAIDs or aspirin within 10 days of study enrollment
* Psychiatric illness or substance abuse that would interfere with ability to comply with protocol requirements or give informed consent
* Surgery within the last 3 months
* Prior gastrointestinal surgery
* Clinically significant infectious, immune mediated or malignant disease
* Receiving an elemental diet or parenteral nutrition
* History of coagulopathy
* Human immunodeficiency virus (HIV) positive
* Hepatitis B surface antigen (HBsAg) positive
* Active cytomegalovirus (CMV)
* Anemia: hemoglobin (Hb) < 8 grams/deciliter (g/dL). If the subject has known significant cardiac disease, subjects with Hb < 10.5 g/dL will be excluded.
* Thrombocytopenia (platelets < 100,000 per microliter [100K/mcL])
* Lymphopenia (absolute lymphocyte count <0.7)
* Immunoglobulin G (IgG) anti-cardiolipin antibody positive >16 International Units (IU)
* Prior exposure to OKT3
* Positive quantiferon gold, tuberculosis (TB) spot test, or purified protein derivative (PPD) test
* Known sensitivity to any ingredients in the study drug
* Anti-mouse antibody titer >1:1000
* Any known autoimmune disease except for ulcerative colitis
* Allergy or hypersensitivity to Omeprazole
* Participated in another clinical trial within 30 days of screening for this trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04-07 (Actual); Primary Completion 2013-05-02 (Actual); Study Completion 2013-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Snapper, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ilan Y, Zigmond E, Lalazar G, Dembinsky A, Ben Ya'acov A, Hemed N, Kasis I, Axelrod E, Zolotarov L, Klein A, El Haj M, Gandhi R, Baecher-Allan C, Wu H, Murugaiyan G, Kivisakk P, Farez MF, Quintana FJ, Khoury SJ, Weiner HL. Oral administration of OKT3 monoclonal antibody to human subjects induces a dose-dependent immunologic effect in T cells and dendritic cells. J Clin Immunol. 2010 Jan;30(1):167-77. doi: 10.1007/s10875-009-9323-7. Epub 2009 Sep 16. PMID 19756989
- [Background] Wu HY, Maron R, Tukpah AM, Weiner HL. Mucosal anti-CD3 monoclonal antibody attenuates collagen-induced arthritis that is associated with induction of LAP+ regulatory T cells and is enhanced by administration of an emulsome-based Th2-skewing adjuvant. J Immunol. 2010 Sep 15;185(6):3401-7. doi: 10.4049/jimmunol.1000836. Epub 2010 Aug 18. PMID 20720210
- [Background] Wu HY, Center EM, Tsokos GC, Weiner HL. Suppression of murine SLE by oral anti-CD3: inducible CD4+CD25-LAP+ regulatory T cells control the expansion of IL-17+ follicular helper T cells. Lupus. 2009 Jun;18(7):586-96. doi: 10.1177/0961203308100511. PMID 19433458
- [Background] Ishikawa H, Ochi H, Chen ML, Frenkel D, Maron R, Weiner HL. Inhibition of autoimmune diabetes by oral administration of anti-CD3 monoclonal antibody. Diabetes. 2007 Aug;56(8):2103-9. doi: 10.2337/db06-1632. Epub 2007 Apr 24. PMID 17456848
- [Background] Ochi H, Abraham M, Ishikawa H, Frenkel D, Yang K, Basso AS, Wu H, Chen ML, Gandhi R, Miller A, Maron R, Weiner HL. Oral CD3-specific antibody suppresses autoimmune encephalomyelitis by inducing CD4+ CD25- LAP+ T cells. Nat Med. 2006 Jun;12(6):627-35. doi: 10.1038/nm1408. Epub 2006 May 21. PMID 16715091

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral OKT3: Participants with ulcerative colitis received 1 milligram (mg) Oral OKT3 given with 20 mg oral Omeprazole once daily for 30 days.
Period: Overall Study
Arm/Group | Oral OKT3
Started | 6
Completed | 4
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: All participants enrolled in the study.
Groups:
- Oral OKT3: Participants with ulcerative colitis received 1 mg Oral OKT3 given with 20 mg oral Omeprazole once daily for 30 days.
Arm/Group | Oral OKT3
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: From baseline to Week 10
Population: All participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral OKT3
Number analyzed (Participants) | 6
Participants | 3

2. Primary Outcome: Number of Participants With Anti-Drug Antibodies
Description: Serum samples were obtained to measure anti-drug antibodies during the study.
Time Frame: From baseline to Week 10
Population: All participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral OKT3
Number analyzed (Participants) | 6
Participants | 0

3. Primary Outcome: Percentage of Biomarker-positive Immune Cells
Description: Peripheral blood mononuclear cells were (PBMCs) were isolated from blood samples taken from each participant at baseline and Week 5. PBMCs were stained with a panel of fluorochrome-conjugated antibodies against multiple surface and intracellular biomarkers, including Cluster of Differentiation (CD) 3, CD4, CD8, Forkhead box P3 protein (FOXP3) and latency-associated peptide (LAP). The percentage of T cells positive for each of these biomarkers was determined by fluorescence activated cell sorting (FACS) and the mean percentage of positive T cells for each biomarker for all analyzed participants is reported.
Time Frame: Baseline, Week 5
Population: All participants enrolled in the study for whom data were available at both time points.
Measure: Mean (Standard Deviation); unit: percentage of biomarker-positive T cells
Arm/Group | Oral OKT3
Number analyzed (Participants) | 6
percentage of biomarker-positive T cells
  CD3, Baseline | 38 (19)
  CD3, Week 5: number analyzed (Participants) | 4
  CD3, Week 5 | 30 (22)
  CD4, Baseline | 59 (30)
  CD4, Week 5: number analyzed (Participants) | 4
  CD4, Week 5 | 75 (11)
  CD8, Baseline | 31 (16)
  CD8, Week 5: number analyzed (Participants) | 4
  CD8, Week 5 | 24 (11)
  FOXP3, Baseline | 5 (2.5)
  FOXP3, Week 5: number analyzed (Participants) | 4
  FOXP3, Week 5 | 4 (2)
  LAP, Baseline | 0.9 (0.5)
  LAP, Week 5: number analyzed (Participants) | 4
  LAP, Week 5 | 0.5 (0.4)

4. Primary Outcome: T Cell Proliferation of PBMCs in Cell Culture
Description: PBMCs isolated from whole blood obtained from participants at baseline, Weeks 1, 3, and 5 were assessed for proliferation in cell culture using a radioactive thymidine incorporation assay. A higher number indicates a higher level of proliferation.
Time Frame: Baseline, Weeks 1, 3 and 5
Population: All participants enrolled in the study for whom data were available at each time point.
Measure: Mean (Standard Error); unit: radioactive counts of cells per minute
Arm/Group | Oral OKT3
Number analyzed (Participants) | 6
radioactive counts of cells per minute
  Baseline | 27470 (12340)
  Week 1 | 49617 (17168)
  Week 3 | 46575 (26762)
  Week 5 | 20993 (15805)

5. Primary Outcome: Cytokine Production by PBMCs in Cell Culture
Description: Cytokine production was assessed in cell cultures of PBMCs obtained from participants at baseline, Weeks 1, 3 and 5. The following cytokines were detected and are reported here: interferon gamma (IFN-gamma), interleukin (IL)-17A, IL-6, IL-1 beta, tumor necrosis factor (TNF) and IL-10.
Time Frame: Baseline, Weeks 1, 3 and 5
Population: All participants enrolled in the study for whom data were available at each time point.
Measure: Mean (Standard Deviation); unit: picograms/milliliter (pg/mL)
Arm/Group | Oral OKT3
Number analyzed (Participants) | 6
picograms/milliliter (pg/mL)
  IFN gamma, Baseline | 4935 (5520)
  IFN gamma, Week 1 | 11521 (6659)
  IFN gamma, Week 3: number analyzed (Participants) | 4
  IFN gamma, Week 3 | 10178 (11671)
  IFN gamma, Week 5: number analyzed (Participants) | 4
  IFN gamma, Week 5 | 2832 (2569)
  IL-17A, Baseline | 69 (93)
  IL-17A, Week 1 | 114 (117)
  IL-17A, Week 3: number analyzed (Participants) | 5
  IL-17A, Week 3 | 181 (368)
  IL-17A, Week 5: number analyzed (Participants) | 4
  IL-17A, Week 5 | 74 (95)
  IL-6, Baseline | 1470 (21010)
  IL-6, Week 1 | 2678 (3270)
  IL-6, Week 3: number analyzed (Participants) | 4
  IL-6, Week 3 | 1978 (3491)
  IL-6, Week 5: number analyzed (Participants) | 4
  IL-6, Week 5 | 567 (57980)
  IL-1 beta, Baseline | 110 (133)
  IL-1 beta, Week 1 | 155 (197)
  IL-1 beta, Week 3: number analyzed (Participants) | 4
  IL-1 beta, Week 3 | 185 (209)
  IL-1 beta, Week 5: number analyzed (Participants) | 4
  IL-1 beta, Week 5 | 38 (30)
  TNF, Baseline | 361 (282)
  TNF, Week 1 | 585 (324)
  TNF, Week 3: number analyzed (Participants) | 3
  TNF, Week 3 | 715 (724)
  TNF, Week 5: number analyzed (Participants) | 4
  TNF, Week 5 | 195 (157)
  IL-10, Baseline | 63 (79)
  IL-10, Week 1 | 115 (124)
  IL-10, Week 3: number analyzed (Participants) | 4
  IL-10, Week 3 | 120 (97)
  IL-10, Week 5: number analyzed (Participants) | 4
  IL-10, Week 5 | 15 (17)

6. Secondary Outcome: Mayo Score
Description: The Mayo Score is determined by the investigator by assigning a score to the following four assessments: stool frequency, rectal bleeding, physician's global assessment and endoscopy. Total range for Mayo score is 0-12 with a higher score indicating a worse outcome.
Time Frame: Baseline, Week 5
Population: All participants enrolled in the study for whom data were available at each time point.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Oral OKT3
Number analyzed (Participants) | 6
score on a scale
  Baseline | 8.8 (1.6)
  Week 5: number analyzed (Participants) | 4
  Week 5 | 7.5 (1.7)

7. Secondary Outcome: Simple Clinical Colitis Activity Index (SCCAI) Score
Description: SCCAI is a symptom based questionnaire addressing five assessments, including bowel frequency day, bowel frequency night, urgency of defecation, blood in stool and general well-being. Score ranges from 0-15 with one additional point added for each manifestation of extracolonic features. A higher score indicates a worse outcome.
Time Frame: Baseline, Week 5
Population: All participants enrolled in the study for whom data were available at each time point.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Oral OKT3
Number analyzed (Participants) | 6
score on a scale
  Baseline | 7.7 (1.6)
  Week 5: number analyzed (Participants) | 4
  Week 5 | 6 (2.5)

8. Secondary Outcome: Score in Histologic Evaluation of Flexible Sigmoidoscopy
Description: Mucosal biopsies were obtained from the most inflamed area seen during flexible sigmoidoscopy and blindly scored by a single pathologist with scores ranging 0-3 with a higher score indicating a worse outcome.
Time Frame: Baseline, Week 5
Population: All participants enrolled in the study for whom data were available at each time point.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Oral OKT3
Number analyzed (Participants) | 6
score on a scale
  Baseline | 2.2 (0.7)
  Week 5: number analyzed (Participants) | 4
  Week 5 | 1.75 (0.9)

ADVERSE EVENTS:
Time Frame: From baseline up to Week 10
Description: The safety population included all participants who received at least one dose of study medication.
Arm/Group | Oral OKT3
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral OKT3 (N=6)
Ulcerative colitis (Gastrointestinal disorders) | 1
Anorectal abscess (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral OKT3 (N=6)
Periorbital edema (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes